CLINICAL TRIAL: NCT05679271
Title: Intracranial Dural Arteriovenous Fistula Related Pulsatile Tinnitus . Endovascular Treatment by Venous Stenting : An Efficacy Study
Brief Title: Dural Sinus Stenting of Low Grade Dural Arteriovenous Fistulae (DAVF) for Pulsatile Tinnitus Treatment
Acronym: INVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: French Ministry of Social Affairs and Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2022/20
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pulsatile Tinnitus
Keywords: Dural arteriovenous fistulae; Pulsatile tinnitus; Venous Stenting
MeSH Terms: conditions — Tinnitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- venous stenting (Experimental): Venous stenting associated to antiaggregation protocol:
  Venous stenting: venous approach can be performed via femoral, brachial or jugular puncture. Autoexpansible stent should delivered at the level of the fistulous sinus. If distal access catheter is wide enough, stent can be delivered directly through it. After partial deployment of the stent, Labbe vein's flow may be restricted. If necessary, several stents can be used in the same procedure to cover the whole length of fistulous sinus area. After stent deployment, ballon angioplasty is compulsory and must be performed using a ballon of equivalent size to the stent. The procedure ends after stent deployment and angiographic arterial post-op controls.
  Antiaggregation protocol: aspirin (160mg for 3 months) + clopidogrel (75mg/d 5 days before stenting and 75mg/d for 1 month after stenting) OR ticagrelor (180mg 2h before stenting and 90mg twice a day for 1 month) in case of clopidogrel platelet resistance.
  Interventions: Device: Venous stenting
- no treatment (Active Comparator): standard care (no treatment)
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Venous stenting — venous stenting associated to antiaggregation protocol
  Arms: venous stenting
Other: Standard of care — observation: no treatment
  Arms: no treatment

SUMMARY:
The goal of this randomized trial to assess the angiographic efficacy of venous stenting in dural arteriovenous fistulae (DAVF) via improvment on Cognard's Classification as compared to no intervention at 6 months Participants belonging to experimental group will be treated using venous stenting. DAVF will be assessed by angiography at 6 months follow-up. Participants belonging to control group will be followed accordingly to standard of care (no treatment). After 6 months, control group patients can be treated by any means accordinlgly to standard of care.

DETAILED DESCRIPTION:
DAVF are frequently revealed as a cause of invalidating pulsatile tinnitus (PT). Endovascular treatment (EVT) of DAVF using liquid embolic agent (LEA) is currently performed when an hemorrhagic risk of intracranial hemorrhage is identified (high grade DAVF). PT alone may not be a sufficient condition to offer EVT because procedure-related risks may overcome clinical benefits specifically in case of extended shunts requiring complex procedures. Stenting of dural sinus may represent an alternative to LEA-EVT with a simple and low risk procedure. Thus PT could be cured even in case of low grade DAVF without neurologic risk.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting invalidating pulsatile tinnitus
* Patient presenting with PT anatomically correlated with a DAVF
* Type I or IIa DAVF on digital subtraction angiography (DSA), according to Cognard's classification.
* DAVF located on sigmoid , lateral or posterior longitudinal sinus.
* Fistula length compatible with use of up to two stents
* Highly effective contraception for women of childbearing potential, maintained during research procedures
* Affiliated or beneficiary of health insurance
* Signed informed consent

Exclusion Criteria:

* Patient with DAVF not eligible for endovascular treatment .
* DAVF classification of IIb or more according to Cognard's classification.
* DAVF with severe sinus stenosis or occlusion judged as nor eligible for sinus stenting.
* DAVF showing evidence of recent (inferior to 3 months) thrombophlebitis at the site of fistulous dural sinus.
* Patient with DAVF previously treated with surgery or radiotherapy.
* Patient with multiple DAVF
* Controlateral sinus aplasia or occlusion
* Patient presenting contra-indication to the use of LEA according to the instructions For Use.
* Patient participating in another clinical study evaluating another medical device,
* Any condition or any situation that would prohibit the patient from coming to the investigational center for the follow-up as recommended by the study protocol at 6 months.
* Patient with any known allergy to heparin, acetylsalicylic acid, Coumadin , Warfarin or other antiplatelet medications
* Patient has undergone a surgery including endovascular procedures in the last 30 days prior to the study procedure.
* Patient has had an Intracranial hemorrhage and/or subarachnoid hemorrhage in the past 30 days prior to the study procedure
* Known serious sensitivity to radiographic contrast agents.
* Known sensitivity to nickel, titanium metals, or their alloys
* Known renal failure as defined by a serum creatinine > 2.5 mg/dl (or 220 μmol/l) or glomerular filtration rate (GFR) < 30.
* Patient who has a contraindication to MRI or angiography for whatever reason
* Women who are pregnant, lactating, or who are planning to become pregnant during the anticipated study period
* Patient unable to understand the nature, risks, significance and implications of the clinical investigation or unwilling to provide written informed consent
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cognard's classification grade | Month 6
  Cognard's classification status : from type I (Anterograde drainage into venous sinus) to Type V (Drainage into the spinal perimedullary veins)

SECONDARY OUTCOMES:
THI score | Baseline, Month 6, Month 12, Month 24
  THI (Tinnitus Handicap Inventory) score (based on 100 points scale from Grade 1 (<16 points) Slight or no handicap to Grade 5 (>=78 points) Catastrophic handicap)
modified Rankin Scale | Baseline, Month 6
  mRS Neurological score (from 0 - No symptoms at all to 6 - Death)
Rate of stent thrombosis | Month 6, Month 12, Month 24
  Rate of stent thrombosis
unsuccessful stent deployment | Baseline
  Rate of unsuccessful stent deployment
Concentration troubles | Baseline, Month 6, Month 12, Month 24
  Assessment via Visual Analog Scale from 0-no trouble to 10-extreme troubles
Sleep troubles | Baseline, Month 6, Month 12, Month 24
  Assessment via Visual Analog Scale from 0-no trouble to 10-extreme troubles
Headaches | Baseline, Month 6
  Assessment via Visual Analog Scale from 0-no trouble to 10-extreme troubles
Dizziness | Baseline, Month 6, Month 12, Month 24
  Assessment via Visual Analog Scale from 0-no trouble to 10-extreme troubles

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No